CLINICAL TRIAL: NCT03767569
Title: Pretreatment With Myo-inositol in Hyperandrogenic PCOS Patients Undergoing ART: a Randomized Controlled Trial
Brief Title: Myo-inositol as Pretreatment in Hyperandrogenic PCOS Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gynositol.2018
Record Dates: First submitted 2018-04-06; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-03

CONDITIONS: PCOS; Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Inositol; Folic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo-inositol (Experimental): Pretreatment with Gynositol (Myo-Inositol 4mg + Folic Acid 0.4mg) daily during 12 weeks before start of ART (Assisted Reproductive Technology)
  Interventions: Drug: Myo-inositol
- Folic acid (Other): Folic acid 0.4 mg daily during 12 weeks before start of ART
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Myo-inositol — Myo-inositol and Folic acid daily
  Arms: Myo-inositol
Drug: Folic Acid — Folic Acid daily
  Arms: Folic acid

SUMMARY:
A randomized controlled trial to evaluate whether pretreatment with myo-inositol can lower testosterone levels and improve clinical outcomes in hyperandrogenic PCOS patients undergoing ART

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* PCOS phenotypes A, B and C
* Signed informed consent

Exclusion Criteria:

* Other relevant endocrine disorders
* Contraindications to the use of gonadotropins
* Endometriosis grade 3-4
* BMI > 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Serum testosterone level after 12 weeks of administration of Myo-Inositol | 2 years

SECONDARY OUTCOMES:
Androstenedione and SHBG (Sex Hormone Binding Globulin) plasma levels after 12 weeks of administration of Myo-Inositol | 2 years
Number of mature oocytes | 2 years
Embryo quality | 2 years
  Day 3 embryos will be classified as transferable or cryopreservable/ 'good-quality embryos' (GQE) according to the criteria described by Van Landuyt et al. (2013). Blastocysts will be categorized according to Gardner et al. (1998) and Gardner and Schoolcraft (1999).
Implantation rate (%) | 2 years
Clinical pregnancy rate (%) | 2 years
Live birth rate in fresh cycle | 2 years
Cumulative live birth rate after 1 cycle | 2 years
Ovarian Hyperstimulation Syndrome rate | 2 years
Consumption of gonadotrophins | 2 years
  measurement in IU
Stimulation days | 2 years
  measurement in days

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided